CLINICAL TRIAL: NCT06724445
Title: Empathy in Frames: Assessing the Impact of Ethnic Concordance in Animated Cartoons on HIV/AIDS Stigma Among South African Young Adults
Brief Title: Empathy in Frames: Animated Cartoons To Reduce HIV Stigma Among South African Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Yanis Ben Amor, Assistant Professor of Global Health and Microbiological Sciences; Executive Director, Center for Sustainable Development in the Climate School, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAU5702
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: HIV-related Stigma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thabo group (Experimental): Participants will view a cartoon video featuring a Black seropositive protagonist
  Interventions: Behavioral: Thabo cartoon
- Steve group (Active Comparator): Participants will view a cartoon video featuring a White seropositive protagonist
  Interventions: Behavioral: Steve cartoon

INTERVENTIONS:
Behavioral: Thabo cartoon — The animated cartoon features Thabo, a Black South African man living with HIV. Through his narrative, viewers follow his daily experiences managing his condition and confronting societal stigma in a South African context. The story explores his interactions with family, friends, and community members, highlighting both challenges and moments of resilience. The animation concludes with Thabo delivering an anti-stigma message directly to viewers.
  Arms: Thabo group
Behavioral: Steve cartoon — The animated cartoon follows Steve, a White man living with HIV. His narrative parallels Thabo's, showing his daily experiences managing HIV and facing societal stigma. The story depicts his interactions with family, friends, and community members, presenting the same situations and challenges as in Thabo's story. The animation ends with Steve delivering the same anti-stigma message to viewers.
  Arms: Steve group

SUMMARY:
This study looks at whether using cartoons that reflect the culture of South Africa can help change how young adults there think about HIV/AIDS. This study will test two types of cartoons in a two-arm (treatment, comparator) randomized controlled trial design-one with Black characters and one with White characters-to see how they affect people's attitudes and knowledge about HIV/AIDS. Randomly allocated participants will be Black seronegative South African adults between 18 and 35 years old. This group was chosen because they're a demographic disproportionately affected by HIV, they're at a high point in their lives for shaping and sharing beliefs, and they're also highly active online, which is where this study takes place.

The cartoons will show the daily struggles of the protagonist living with HIV/AIDS, and end with a call to action. The study aims to highlight how the characters' ethnicity influences how viewers feel about and remember the message. The investigators want to understand if seeing characters who look like them helps people understand and empathize more. The aim of this study is to learn how cultural representation can improve health communication and guide future efforts to reduce stigma in different communities. Ultimately, the investigators hope this study will contribute to better public health messages and create a more accepting environment for people with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Must self-identify as Black South African
* Must be HIV seronegative
* Age range: 18-35 years
* Must currently reside in South Africa
* Must have basic English language comprehension
* Must have internet access to view video content

Exclusion Criteria:

* Prior participation in HIV stigma reduction interventions
* HIV seropositive status
* Non-Black South African identity
* Outside target age range (18-35)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1496 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Attitudes towards HIV | Up to 14 days
  HIV-related attitudes are measured using Beaulieu et al's SAT-PLWHA-S survey instrument, designed specifically to measure stigmatizing attitudes towards HIV/AIDS. The objective of this questionnaire is to measure participants' own HIV-related behaviors. This measurement uses a 5-point Likert-type scale (from 1 =strongly disagree to 5 = strongly agree) to understand how participants behave when confronted with HIV-related information. Respondents will be asked to answer items such as "Stories featuring diverse ethnic backgrounds make me feel more connected to the content" or "Ethnic diversity in health messages affects my trust in their accuracy".
  A higher score indicates more positive attitudes and comfort levels regarding HIV and people living with HIV.
Health Ethnicity Perceptions | Up to 14 days
  A composite index measuring participants' perceptions of the relevance, relatability, and trustworthiness of health messages based on the ethnicity of the message source. Items assess how protagonist ethnicity influenced viewers' ability to engage with the content, trust the information, and find the message relatable.
  3-item Likert scale index (1-5), with higher scores indicating more positive perceptions of ethnic concordance in health messaging.

SECONDARY OUTCOMES:
Behavioral intentions | Up to 14 days
  Behavioral Intentions will be measured using a shortened version of the Theory of Planned Behavior (TPB) Questionnaire used to assess attitudes toward the behavior, subjective norms, and perceived behavioral control. Focusing on attitudes, subjective norms, perceived behavioral control, and intention towards a specific behavior (e.g., engaging in HIV prevention practices) can yield a concise measure. This measure uses a 5 point Likert-type scale (from 1 = strongly disagree to 5 = strongly agree).
  A higher score indicates greater readiness and confidence to engage in HIV stigma reduction activities.
HIV knowledge | Up to 14 days
  HIV knowledge is assessed using a shortened version of Carey and Colls' HIV Knowledge Questionnaire (HIV-KQ-18). Respondents will be required to rate their understanding of the infection, transmission, and treatment of HIV on a binary scale (1 = true, 2 = false). Typical questions range from "Can HIV be transmitted by sharing food with someone who is HIV positive?" to "A person with HIV can have an undetectable viral load with proper treatment".
  A higher score indicates greater certainty of HIV knowledge.
Viewer Engagement with Cartoon | 14 days
  Quality of engagement will be measured using a shortened version of the User Engagement Scale (UES) adapted for health-related animated cartoons. This scale is designed to provide insights into how these interventions capture and hold the audience's attention, and potentially influence their health knowledge and behaviors. This measurement uses a 5-point Likert-type scale (from 1 = strongly disagree to 5 = strongly agree) to measure focused attention, perceived usability, aesthetic appeal, reward, and endurability.
  A higher score indicates greater perceived effectiveness and engagement with cartoon-based HIV health messaging.

CONTACTS AND LOCATIONS:
Overall Officials: Yanis Ben Amor, PhD, Study Chair — Columbia University; Adam Sacarny, PhD, Study Chair — Columbia University
Locations (1):
- Busara Center for Behavioral Economics, Multiple Locations, South Africa

IPD SHARING:
Plan to Share IPD: No